CLINICAL TRIAL: NCT01746771
Title: A Phase I-II Study to Assess the Safety, Efficacy and Pharmacokinetic Profile of HM781-36B Combined With Paclitaxel and Trastuzumab in Patients With HER-2 Positive Advanced Gastric Cancer
Brief Title: A Phase I-II Study of HM781-36B Combined With Paclitaxel and Trastuzumab in HER-2 Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: National OncoVenture (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-PHI-A201
Record Dates: First submitted 2012-12-03; First posted 2012-12-11 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: HER-2 Positive Advanced Gastric Cancer
Keywords: HM781-36B, Paclitaxel, Trastuzumab
MeSH Terms: interventions — HM781-36B; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM781-36B, Paclitaxel, Trastuzumab (Experimental): HM781-36B(Poziotinib): QD*2weeks/3weeks Paclitaxel: 175mg/m2 Trastuzumab(Herceptin): 8mg/kg
  Interventions: Drug: HM781-36B(Poziotinib); Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: HM781-36B(Poziotinib) — QD*2weeks/3weeks
  Other Names: NOV120101; Poziotinib
Drug: Paclitaxel — 175mg/m2
Drug: Trastuzumab — 8mg/kg
  Other Names: Herceptin

SUMMARY:
[Phase I] The main objective of this study is to evaluate the safety, tolerability and determine the Recommended Dose (RD) of HM781-36B(Poziotinib)combined with Paclitaxel and Trastuzumab

[Phase II] The main objective of this study is to evaluate anticancer activity through determination of response rate of HM781-36B(Poziotinib)combined with Paclitaxel and Trastuzumab in patients with HER-2 positive advanced gastric cancer

DETAILED DESCRIPTION:
Besides the main objectives, there are other objectives as follows:

[Phase I]

1. To assess the pharmacokinetic profile of HM781-36B(Poziotinib) combined with Paclitaxel and Trastuzumab
2. To evaluate anticancer activity of HM781-36B(Poziotinib) combined with Paclitaxel and Trastuzumab in patients with HER-2 positive advanced gastric cancer
3. To evaluate PFS(Progression-Free Survival), TTP (Time To Tumor Progression), and DOR (Duration of Overall Response)

[Phase II]

1. To assess the safety, tolerability of HM781-36B(Poziotinib) combined with Paclitaxel and Trastuzumab
2. To evaluate tumor response through determination of disease control rate , PFS(Progression-Free Survival), TTP (Time To Tumor Progression), and DOR (Duration of Overall Response)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced gastric cancer including gastroesophageal junction adenocarcinoma
2. At least one measurable lesion defined by RECIST(v1.1)
3. FISH+ or IHC3+ (regardless of FISH results)
4. Age≥19
5. ECOG ≤ 2
6. Life expectancy ≥ 12 weeks
7. Adequate bone marrow and no abnormal heart and lung function
8. No radiotherapy, other anticancer drugs or immunotherapy is allowed during this study
9. Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up assessments and procedures

Exclusion Criteria:

1. Patients with a history of hypersensitivity to Trastuzumab and who have been treated with medicine including Cremophor EL
2. Patients who have a current active malignancy other than gastric adenocarcinoma (with exception of non-melanoma skin cancer or cervical cancer in situ)
3. Patients who have previously received taxane-based chemotherapy
4. The presence of central nervous system metastases
5. Patients who have a blood tumor such as leukemia, or who had previously received, or are planning to receive, the bone marrow transplant
6. Patients with uncontrolled infection
7. Patients who have GI malabsorption or difficulty taking oral medication
8. Patients with following diseases are excluded:
9. Patients with psychiatric or congenital disorder which can affect adherence or make hard to follow the requirements of the protocol
10. Pregnant or breastfeeding women or women of childbearing who do not use an appropriate method of contraception (male patient should also use an appropriate method of contraception)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety evaluation(phase I) | DLT will be evaluated on Day 21 during cycle 1
  Dose limiting toxicity (DLT), Maximum tolerance dose (MTD)

SECONDARY OUTCOMES:
Efficacy evaluation(Phase II) | Efficacy will be evaluated every 6 weeks or 9 weeks
  Efficacy evaluation; phase II (Simon's two-stage minimax design): Disease Control Rate (CR, PR, SD), PFS(Progression-Free Survival), TTP (Time To Tumor Progression), and DOR (Duration of Overall Response)

CONTACTS AND LOCATIONS:
Overall Officials: YoHan Kim, M.D., Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- Seoul National University Hospital, Seoul, South Korea